CLINICAL TRIAL: NCT01562899
Title: A Phase Ib/II Open-label, Multi-center Study of the Combination of MEK162 Plus AMG 479 (Ganitumab) in Adult Patients With Selected Advanced Solid Tumors
Brief Title: A Study of MEK162 and AMG 479 in Patients With Selected Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was withdrawn due to scientific and business considerations.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CMEK162X2111; C4211010 (Other: Alias Study Number); 2012-000305-76 (EudraCT Number)
Record Dates: First submitted 2012-03-22; First posted 2012-03-26 (Estimated); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Metastatic Pancreatic Adenocarcinoma; BRAF Mutated Melanoma
Keywords: MEK162; AMG 479; Ganitumab; colorectal adenocarcinoma; pancreatic adenocarcinoma; melanoma; KRAS; BRAF
MeSH Terms: conditions — Melanoma | interventions — binimetinib; ganitumab

ARMS (4):
- Dose escalation (Experimental): Dose finding group chosen in order to establish a safe and tolerated dose of binimetinib in combination with ganitumab in patients with selected advanced solid tumors.
  Interventions: Drug: MEK162; Drug: AMG 479
- KRAS mutated colorectal adenocarcinoma (Experimental): Patients with KRAS mutant colorectal cancer.
  The starting dose (30 mg bid) of binimetinib chosen for this study was a fraction of the MTD (60 mg bid) and the RP2D (45 mg bid) determined for single agent use. The starting dose for ganitumab was 12 mg/kg q2w which had been shown to be a well-tolerated dose in combination with other anti-cancer agents.
  Interventions: Drug: MEK162; Drug: AMG 479
- Metastatic pancreatic adenocarcinoma (Experimental): Patients with metastatic pancreatic cancer.
  The starting dose (30 mg bid) of binimetinib chosen for this study was a fraction of the MTD (60 mg bid) and the RP2D (45 mg bid) determined for single agent use. The starting dose for ganitumab was 12 mg/kg q2w which had been shown to be a well-tolerated dose in combination with other anti-cancer agents.
  Interventions: Drug: MEK162; Drug: AMG 479
- BRAF mutated melanoma (Experimental): Patients with mutant BRAF V600 melanoma.
  The starting dose (30 mg bid) of binimetinib chosen for this study was a fraction of the MTD (60 mg bid) and the RP2D (45 mg bid) determined for single agent use. The starting dose for ganitumab was 12 mg/kg q2w which had been shown to be a well-tolerated dose in combination with other anti-cancer agents.
  Interventions: Drug: MEK162; Drug: AMG 479

INTERVENTIONS:
Drug: MEK162 — Supplied as tablets of dosage strength 15 mg in high-density polyethylene bottles with child-resistant closure.
  Other Names: Binimetinib
Drug: AMG 479 — Supplied as sterile liquid for intravenous infusion in vials in boxes. Until April 2013 a frozen formulation with a concentration of 30 mg/ml was used; from May 2013 onwards a refrigerated formulation with a concentration of 70 mg/ml was used.
  Other Names: Ganitumab

SUMMARY:
This is a multi-center, open-label, phase Ib/II study. First, the aim of the phase Ib part is to estimate the MTD(s) and/or to identify the recommended phase II dose(s) (RP2D) for the combination of MEK162 and AMG 479 (ganitumab), followed by the phase II part to assess the clinical efficacy and to further assess the safety of the combination in selected patient populations. The dose escalation part of the study will be guided by a Bayesian Logistic Regression Model (BLRM). At least 18 patients are expected to be enrolled in the dose escalation part.

Following MTD/ RP2D declaration, patients will be enrolled in three phase II arms to assess efficacy of the combination as well as to better understand the safety, tolerability, PK, antibody concentrations and PD of the combination at MTD/RP2D. Phase II arm 1 will consist of approximately 25 patients with KRAS-mutant colorectal adenocarcinoma. Phase II arm 2 will consist of approximately 20 patients with metastatic pancreatic adenocarcinoma. Phase II arm 3 will consist of approximately 28 patients with mutant BRAFV600 melanoma.

Patients will be treated until progression of disease, unacceptable toxicity develops, or withdrawal of informed consent, whichever occurs first. All patients will be followed up - at minimum patients must complete the safety follow-up assessments 30 days after the last dose of the study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years
* Patients with advanced solid tumors (CRC, melanoma) with documented somatic KRAS or BRAFV600 mutations in tumor tissue. Patients with metastatic pancreatic adenocarcinoma may be enrolled irrespectively of KRAS or BRAFV600 mutational status.
* Patients must have relapsed or progressed following standard therapy or patients for whom no standard anticancer therapy exists.
* Measurable disease as determined by RECIST v1.1. World Health Organization (WHO) Performance Status (PS) ≤ 2.
* Adequate organ function
* Negative serum pregnancy test

Exclusion Criteria:

* Prior therapy with MEK- or IGF-1R- inhibitor
* History or current evidence of central serous retinopathy (CSR), retinal vein occlusion (RVO) or retinal degenerative disease
* Patients with known history of severe infusion reactions to monoclonal antibodies
* Patients with primary CNS tumor or CNS tumor involvement
* History of thromboembolic event requiring full-dose anticoagulation therapy
* Clinically significant cardiac disease
* History of another malignancy within 2 years
* Pregnant or nursing (lactating) women

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2012-08-27 (Actual); Primary Completion 2015-04-01 (Actual); Study Completion 2015-04-01 (Actual)

PRIMARY OUTCOMES:
Phase Ib: Estimation of Maximum Tolerated Doses (MTDs) and/or recommended Phase II doses (RP2Ds) by measuring incidence of dose limiting toxicities | Approximately 6 months
  To estimate the MTDs and/or RP2Ds of MEK162 in combination with AMG479 by measuring incidence of dose limiting toxicities in Cycle 1 (Cycle 1 = 28 days)
Phase II: Antitumor activity of MEK162 in combination with AMG 479 by evaluating Objective Response Rate (ORR) in colorectal carcinoma and melanoma and by evaluating Disease Control Rate (DCR) at week 10 in pancreatic carcinoma | Approximately 24 months
  To estimate the antitumor activity of MEK162 in combination with AMG479 by evaluating Objective Response Rate (ORR) according to RECIST 1.1 in colorectal carcinoma and melanoma and by evaluating the Disease Control Rate (DCR) per RECIST 1.1 at week 10 in pancreatic carcinoma

SECONDARY OUTCOMES:
Both Phases: Safety and tolerability of MEK162 & AMG 479 (ganitumab) in combination by evaluating the adverse events, serious adverse events, changes in hematology and chemistry values, vital signs, ECGs; dose interruptions, reductions and dose intensity | Phase Ib: Approximately 6 months; Phase II: Approximately 24 months
  To characterize the safety and tolerability of MEK162 and AMG 479 (ganitumab) in combination by evaluating the incidence and severity of adverse events, serious adverse events (as per CTCAE grading), changes in hematology and chemistry values, vital signs, ECGs; dose interruptions, reductions and dose intensity
Both Phases: Determination of single and multiple dose pharmacokinetics (PK) profile of MEK162 in combination with AMG 479 (ganitumab) by measuring time vs. plasma concentrations and basic PK parameters of MEK162 | Phase Ib: Approximately 6 months; Phase II: Approximately 24 months
  To determine single and multiple dose PK profile of MEK162 in combination with AMG 479 (ganitumab) by measuring time vs. plasma concentration as well as basic PK parameters of MEK162 at different timepoints prior and post study drug combination dosing.
Phase Ib: Preliminary anti-tumor activity of MEK162 and AMG 479 (ganitumab) in combination by evaluating the Overall Response Rate (ORR), Duration of Response (DOR) and Progression Free Survival (PFS) | Approximately 6 months
  To assess preliminary anti-tumor activity of MEK162 and AMG 479 (ganitumab) in combination by evaluating Overall Response Rate (ORR), Duration of Response (DOR), Progression Free Survival (PFS) as assessed by the investigator according to RECIST 1.1
Phase II: Further anti-tumor activity of MEK162 & AMG 479 (ganitumab) in combination by evaluating the DOR, PFS and OS by evaluating Disease Control Rate for colorectal carcinoma and melanoma; Overall Response Rate for pancreatic carcinoma patients | Approximately 24 months
  To further assess the anti-tumor activity of MEK162 and AMG 479 (ganitumab) in combination by evaluating the Duration of Response (DOR) and Progression Free Survival (PFS) per RECIST 1.1 and Overall Survival in all phase II patients and by evaluating the Disease Control Rate (DCR) per RECIST 1.1 for colorectal carcinoma and melanoma and Overall Response Rate (ORR) per RECIST 1.1 for pancreatic carcinoma patients

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- United States (2):
  - Massachusetts General Hospital Mass General 2, Boston, Massachusetts
  - University of Utah / Huntsman Cancer Institute Huntsman, Salt Lake City, Utah
- Pfizer Investigative Site, Parkville, Victoria, Australia
- Pfizer Investigative Site, Leuven, Belgium
- Pfizer Investigative Site, Toronto, Ontario, Canada
- Pfizer Investigative Site, Toulouse, France
- Pfizer Investigative Site, Napoli, Italy
- Pfizer Investigative Site, Barcelona, Catalonia, Spain
- Pfizer Investigative Site, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests